CLINICAL TRIAL: NCT00460863
Title: Effects of Hemodialysis on the Slee/Wake Cycle of Patients on Chronic Hemodialysis
Brief Title: Effects of Hemodialysis on the Sleep/Wake Cycle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sandra B. Dunbar, RN, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0602-2002; R01NR004340 (NIH); 72728732 (Other: Other)
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2008-05

CONDITIONS: End Stage Renal Disease
Keywords: sleep; hemodialysis; daytime sleepiness; temperature
MeSH Terms: conditions — Kidney Failure, Chronic; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: using cool versus warm dialysate during hemodialysis

SUMMARY:
The purpose of this study is to test a novel application of an existing treatment - using col dialysate (often used to treat hypotension) as opposed to warm dialysate (standard treatment) during hemodialysis for its ability to stabilize the sleep/wake cycle of patients receiving this chronic treatment

DETAILED DESCRIPTION:
This competing continuation proposal follows NR04340, "The Effects of Hemodialysis on the Sleep/ Wake Cycle", and seeks to test the efficacy of altering dialysate temperature on nocturnal sleep and daytime sleepiness in patients on chronic hemodialysis (HD). During the initial funding period, we examined the effects of HD and the time of its administration on sleep and waking. The major findings were that, in comparison to a group of control subjects with renal failure not yet on dialysis, HD subjects had reduced nocturnal total sleep time and sleep efficiency and increased numbers of brief arousals. One-third of HD subjects had abnormal, objectively measured daytime sleepiness, significant predictors of which were indices of nocturnal sleep disorders and duration of HD treatment. These effects occurred independent of treatment time of day. The negative influence of daytime sleepiness on life quality and functioning that we also found highlights the importance of the development and testing of interventions designed to address these changes. Furthermore, the recently described relationship between sleep disorders/sleepiness and cardiovascular disease leading cause of death in HD patients underscores the importance of this work.

Within the context of the Two-Process Model of Sleep Regulation and the well-described relationship between sleep/wake state and body temperature (BT), the data from additional studies we have conducted indicate that HD associated heat production contributes to its iatrogenic effects on the sleep/wake cycle. Consistent with other reports, we have shown that HD causes an increase in BT and, furthermore, alters its course across the day. We have also shown that BT and state sleepiness predictably covary across the duration of HD and that HD is associated with increased levels of both subjective and objective measurements of sleepiness. From both theoretical and physiological perspectives, one would predict that these HD-induced changes would place patients at high-risk for sleep/wake disturbances. In fact, both the nocturnal and daytime polysomnographic studies we conducted during our initial funding period demonstrate the severity of the sleep/wake problems experienced by this group. Previously tested interventions designed to improve the sleep of HD patients, such as normalizing hematocrit and performing slow, nocturnal HD, have decreased periodic limb movements and sleep apnea respectively, but have failed to significantly improve other indices of nocturnal sleep quality. We thus conducted a pilot study to test our hypothesis that treatment induced changes in BT contribute to the fragmented nocturnal sleep seen in this group by using cool dialysate (an existing intervention used to reduce hypotension) to block heat production and stabilize the sleep/wake cycle. Preliminary results demonstrated that, after one treatment, this intervention markedly normalized the rhythm of BT and improved indices of nocturnal sleep quantity and quality. Therefore, a major component of this proposal is to test a novel application for a safe, non-pharmacologic, cost-effective intervention that is already in use in clinical practice - using cool dialysate during HD to help stabilize the sleep/wake cycle of chronic HD patients. We will also evaluate its effects on selected sleep-related physiologic, psychological, behavioral, and general health outcomes.

This study, a randomized, single-blinded, control group clinical trial, represents the logical progression of a program of research devoted to the development of interventions designed to optimize the sleep/wake patterns of patients on chronic HD. The specific aims and associated hypotheses are:

1. To test the effects of using cool dialysate during HD in comparison to warm dialysate (standard treatment) on the sleep/wake cycle of patients with chronic renal failure.

   H1 HD subjects will have improved nocturnal sleep (objective and subjective measures of sleep latency, total sleep time, sleep efficiency, and sleep disturbance) when dialyzed with cool dialysate in comparison to a warm dialysate.

   H2 HD subjects will have decreased daytime sleepiness (physiologic, manifest, and introspective) when dialyzed with cool dialysate in comparison to warm dialysate .
2. To test the effects of using cool dialysate during HD in comparison to warm dialysate on other sleep-related physiological, psychological, behavioral, and general health outcomes.

H3 HD subjects will demonstrate improvement in selected sleep-related physiological (distal/proximal skin gradient and axillary body temperature rhythm), psychological (mood), behavioral (daily rest/activity), and general health outcomes (quality of life and functional status) when dialyzed with cool dialysate in comparison to warm dialysate.

ELIGIBILITY:
Inclusion Criteria:

* All races
* Cause of renal failures - diabetes, hypertension, glomerulonephritis, or polycystic kidney disease
* Ability to read and write in English hemodialysis three times a week for at least 4 months
* Clinically stable
* KT/V > 1.0

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Polysomnographic measures of sleep | At three time points over the nine month study period
Polysomnographic measures of daytime sleepiness | At three time points over the nine month study period
Distal/proximal skin temperature gradient | At three time points during the nine month study period

SECONDARY OUTCOMES:
Subjective measure of sleep quality | Monthly during the nine month study period
Subjective measure of daytime sleepiness | Monthly during the nine month study period
Subjective measure of mood | Monthly during the nine month study period
Subjective measure of quality of life | Monthly during the nine month study period
Subjective measure of functional health status | Monthly during the nine month study period

CONTACTS AND LOCATIONS:
Overall Officials: Kathy P Parker, PhD, Principal Investigator — Emory University
Locations (1):
- Nell Hodgson Woodruff School of Nursing, Atlanta, Georgia, United States